CLINICAL TRIAL: NCT04860362
Title: Effectiveness of a Telehealth Group for Improving Peer Relationships for Adolescents With Neurofibromatosis Type 1
Brief Title: Pilot Randomized Control Trial of Telehealth Group for Improving Peer Relationships (PEERS) in NF1
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Wisconsin, Milwaukee (Other)
Collaborators: NF Midwest (Unknown); NF Northeast (Unknown)
Responsible Party: Principal Investigator, Bonita P Klein-Tasman, Professor, University of Wisconsin, Milwaukee
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 21-039-UWM-b
Record Dates: First submitted 2021-04-19; First posted 2021-04-26 (Actual); Last update posted 2021-04-26 (Actual); Status verified 2021-04

CONDITIONS: Neurofibromatosis 1; Social Skills
MeSH Terms: conditions — Neurofibromatosis 1; Social Skills

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): PEERS weekly sessions - parallel teens and parent/caregiver groups
  Interventions: Behavioral: PEERS
- Wait List Control (Other): Offered intervention at a later date
  Interventions: Behavioral: PEERS

INTERVENTIONS:
Behavioral: PEERS — Structured social skills curriculum including didactics, behavioral rehearsal, parent coaching, and parent coaching support.
  Other Names: Program for the Education and Enrichment of Relational Skills

SUMMARY:
This is a pilot randomized control trial of the UCLA PEERS protocol delivered via Telehealth with teens with neurofibromatosis type 1 whose parents report that they have difficulty making and keeping friends.

ELIGIBILITY:
Inclusion Criteria:

* Physician diagnosis of neurofibromatosis type 1
* Age 12-17
* Main language spoken in the home is English
* Reliable internet access
* Current functional impairment in peer relationships
* Teen is interested and motivated to participate

Exclusion Criteria:

* Main language spoken in the home is not English
* Cognitive or developmental difficulties that affect reading comprehension or understanding of treatment material
* Significant behavioral concerns
* Other comorbid medical conditions
* Major surgery in past 6 months
* Prior social skills group treatment within past 6 months
* Prior participation in PEERS

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2021-01-29 (Actual); Primary Completion 2021-09 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
Social Skills Improvement System - SEL (SSIS-SEL; Gresham & Elliot, 2017) Parent | within 4 weeks of PEERS completion
  Change from pre- to post-test on SSIS-SEL parent Total Standard Score (measures social functioning)
Test of Adolescent Social SKills (TASSK: Laugeson & Frankel, 2010) | within four weeks of PEERS completion
  Change from pre- to post-test on total score (measures knowledge of the PEERS concepts)
Social Skills Improvement System - SEL (SSIS-SEL; Gresham & Elliot, 2017) Parent | 16 weeks following PEERS completion
  Change from pre- to 16 week followup on total score
Social Skills Improvement System - SEL (SSIS-SEL; Gresham & Elliot, 2017) Parent | within four weeks of PEERS completion for treatment group
  Amount of change from pre- to post-test differs from change in Wait List Control group

SECONDARY OUTCOMES:
Social Responsiveness Scale -2 (SRS-2; Constantino, 2005) | within 4 weeks following PEERS completion
  change from pre- to post-test on Total SRS-2 completed by caregivers (measure of social impairment)
Social Responsiveness Scale -2 (SRS-2; Constantino, 2005) | 16 weeks following PEERS completion
  change from pre- to 16 week followup on Total SRS-2 completed by caregivers (measure of social impairment)
Social Skills Improvement System - SEL (SSIS-SEL; Gresham & Elliot, 2017) Teen | within 4 weeks of PEERS completion
  Change from pre- to post-test on teen self-report of social functioning
Social Skills Improvement System - SEL (SSIS-SEL; Gresham & Elliot, 2017) Teen | 16 weeks following PEERS completion
  Change from pre- to 16 week followup on teen self-report of social functioning

OTHER OUTCOMES:
Peds QL (Varni et al, 2002) Parent | within 4 weeks of PEERS completion
  Change from pre- to post-test in parental ratings of QoL
Peds QL (Varni et al, 2002) Teen | within 4 weeks of PEERS completion
  Change from pre- to post-test in teen ratings of QoL

CONTACTS AND LOCATIONS:
Overall Officials: Bonnie Klein-Tasman, PhD, Principal Investigator — University of Wisconsin, Milwaukee
Locations (1):
- University of Wisconsin-Milwaukee, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data will be available upon request to qualified investigators.
Supporting Information: Study Protocol, ICF
Time Frame: Available following publication of the research study.
Access Criteria: Contact the PI (bklein@uwm.edu)